CLINICAL TRIAL: NCT06195774
Title: Impact on Respiratory Function Associated to Epidural Analgesia in Parturient Women as Assessed by Electrical Impedance Tomography: a Monocentric Prospective Study
Brief Title: Effect of Epidural Analgesia on Regional Lung Ventilation in Parturient Women as Assessed by Thoracic Impedance
Status: Not yet recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2023422
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Complications; Atelectasis
Keywords: pregnancy; labor; at term; electric impedance tomography; pulmonary impedance
MeSH Terms: conditions — Pregnancy Complications; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: Measure regional electric impedance of the lung for before and after insertion of an epidural analgesia catheter

SUMMARY:
The goal of this observational study is to learn more about the effect of obstetric epidural anesthesia on regional lung ventilation in healthy parturient women. The main question it aims to answer is whether the initiation or epidural analgesia improves or not regional lung ventilation in healthy women at term during labor.

Participants will be subject to measurements of pulmonary impedance by electric impedance tomography before and after the start of epidural analgesia. No change will be applied to clinical care as a result of this measurement.

ELIGIBILITY:
Inclusion Criteria:

* At-term pregnancy (at least 36 weeks)
* ASA class I-II

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) Class III or more
* BMI>35 before pregnancy
* Contraindication to routinely administrated drugs (levobupivacaine, lidocaine, sufentanil)
* Contraindication to epidural analgesia
* Pregnancy-related complications (including pre-eclampsia)
* Respiratory system diseases
* Severe psychiatric disorders
* Twin pregnancy
* Skin lesions in correspondence to the position of the Electric impedance tomography belt
* Pacemaker or Implantable Cardioverter Defibrillator (ICD)
* Language barrier

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include healthy pregnant patients that come for spontaneous or induced labor at the hospital's delivery room.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Regional lung ventilation (ROI 1-4) | "before" measurements will be taken just before applying lumbar epidural analgesia, and "after" measurements will be taken 5 minutes and ten minutes after starting lumbar epidural analgesia. Measurements take 10 minutes of continuous registration
  Assess regional ventilation as measured by electric impedance in each of the 4 Regions Of Interest (from anterior to posterior) in which the lung is divided, before and after epidural analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Szegedi, M.D., Ph.D., Principal Investigator — Erasmus University Hospital
Locations (1):
- Erasmus University Hospital, Brussels, Anderlecht, Belgium

IPD SHARING:
Plan to Share IPD: Undecided